CLINICAL TRIAL: NCT03712618
Title: Short or Long Infusion Duration for Platelets: The SOLID Platelet Study
Brief Title: The SOLID Platelet Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to recruitment difficulty
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 190005; 19-CC-0005
Record Dates: First submitted 2018-10-18; First posted 2018-10-19 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-02

CONDITIONS: Platelet Transfusion Refractoriness (PTR); Thrombocytopenia
Keywords: Platelet Transfusion Refractoriness; Continuous Platelet Transfusion
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A: LONG then SHORT transfusion (Active Comparator): Subjects with thrombocytopenia (due to congenital causes, bone marrow failure, hematologic malignancies, and treatment-related) randomized to receive LONG platelet transfusion (Transfused over 4-HOURS via infusion pump or gravity) with follow up until 6 hours and then SHORT platelet transfusion (Transfused over 60-minutes via infusion pump or gravity) with follow up until 6 hours for a combined total of 12 hours. Subjects may receive up to two further subsequent blocks (one per day) to be administered to a subject in alternating order of SHORT and LONG platelet transfusions, for a maximum number of three blocks per subject.
  Interventions: Biological: Platelet Transfusion - LONG Platelet Transfusion; Biological: Platelet Transfusion - SHORT Platelet Transfusion
- Group B: SHORT then LONG transfusion (Active Comparator): Subjects with thrombocytopenia (due to congenital causes, bone marrow failure, hematologic malignancies, and treatment-related) randomized to receive SHORT platelet transfusion (Transfused over 60-minutes via infusion pump or gravity) with follow up until 6 hours and then LONG platelet transfusion (Transfused over 4-HOURS via infusion pump or gravity) with follow up until 6 hours for a combined total of 12 hours. Subjects may receive up to two further subsequent blocks (one per day) to be administered to a subject in alternating order of LONG and SHORT platelet transfusions, for a maximum number of three blocks per subject.
  Interventions: Biological: Platelet Transfusion - LONG Platelet Transfusion; Biological: Platelet Transfusion - SHORT Platelet Transfusion

INTERVENTIONS:
Biological: Platelet Transfusion - LONG Platelet Transfusion — Platelets transfused over 4-HOURS
Biological: Platelet Transfusion - SHORT Platelet Transfusion — Platelets transfused over 60-minutes

SUMMARY:
Background:

Platelets are cell fragments in the blood that help it clot. Some people get very low platelet counts during a disease or treatment. Low platelet counts can cause severe bleeding. Some people are not helped by platelet transfusions at the standard transfusion rate. This is called platelet transfusion refractoriness (PTR). Researchers want to learn more about transfusing platelets so they can make transfusions more effective.

Objectives:

To study the effects of transfusing platelets more slowly than the standard rate. To obtain data to improve the effectiveness of platelet transfusions in people with PTR and decrease the risk of bleeding in some people.

Eligibility:

Adults ages 18-100 who have very low platelet counts requiring platelet transfusion, and have evidence of PTR

Design:

Participants will be screened with a review their recent NIH medical records. They will have blood drawn.

Participants will have up to three 12-hour treatment blocks. They can have only one block per day. During each block, they will have 2 platelet transfusions in those 12 hours.

One transfusion will take place over 1 hour (SHORT infusion). The other will take place over 4 hours (LONG infusion).

Participants will be randomly put in 1 of 2 treatment groups. This will dictate whether they get the SHORT or LONG infusion first.

Participants will have blood drawn:

* When they enroll
* Right before each transfusion
* 2, 4, and 6 hours after each transfusion

Each blood draw will consist of a complete blood count. Smaller tubes that require only small amounts of blood will be used to minimize the amount of blood drawn.

DETAILED DESCRIPTION:
Platelet transfusion can be a life-saving procedure in preventing or treating serious bleeding in patients who have low and/or dysfunctional platelets. Treatment of blood cancer and other blood diseases, as well as bone marrow transplantation, is not possible without platelet transfusion support. Unfortunately, 15- 25% of chronically transfused patients platelet counts will stop responding to these transfusions, putting them at risk for serious bleeding complications. The development of human leukocyte antigen (HLA) antibodies is responsible for 4- 8% of this platelet transfusion refractoriness. The presence of HLA antibodies is a clinical complication that is generally managed by the selection of products that are negative for the antigens for which the patient has antibodies. Often, for patients with chronic and ongoing need, this selection is facilitated by targeted recruitment of donors with known HLA types (i.e., types that lack antigens cognate to the patients known antibodies and are thus predicted to be compatible). However, for very broadly HLA- alloimmunized patients, compatible products may be exceedingly scarce or completely unavailable, precluding the ability to consistently provide products the patient will likely increment from. This research protocol is designed to evaluate the efficacy of a 4-hour continuous infusion of single donor, apheresis platelets in overcoming both alloimmune-mediated and non-alloimmune-mediated platelet refractoriness. We hypothesize that when we transfuse patients over a long duration, who have platelet refractoriness, the platelet counts will increase to higher numbers for an extended period of time in the peri-transfusion period when compared to shorter transfusion intervals.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Ability to comprehend the investigational nature of the study and provide informed consent
* Thrombocytopenia

  * Causes of thrombocytopenia may be due to:

    1. Congenital causes
    2. Bone marrow
    3. Hematologic malignancies
    4. Treatment related
  * Thrombocytopenia is generally defined as one of the following:

    1. Platelet count <10K/uL without bleeding
    2. Platelet count <20K/uL for "complicated prophylaxis" in patients determined to be at increased risk of bleeding or other complications
    3. Platelet count <50K/uL with evidence of active bleeding, such as intracranial hemorrhage, GI bleeding, pulmonary hemorrhage, uncontrolled epistaxis, hematuria.

       The treating provider may change the platelet transfusion threshold based on the clinical circumstance, patient population, and/or concurrent primary protocol considerations - similar to the PLADO study.
* Diagnosed with PTR, characterized by the following:

  * Lack of adequate post-transfusion platelet count increment, defined by, Corrected Count Increment (CCI) <5000/ul at 10-60 min after each of at least 2 consecutive platelet transfusions
  * Presence of anti-HLA class 1 type A and/or type B antibody, in the setting of PTR, as defined above, constitutes the HLA alloimmune-mediated subtype of PTR. Presence of one or more HPA antibodies in the setting of PTR, as defined above, constitutes the HPA alloimmune-mediated subtype of PTR. Failure to detect HLA or HPA antibodies will be categorized as non-alloimmune-mediated PTR. .

EXCLUSION CRITERIA:

* Less than 18-years-old
* Lack of ability to obtain informed consent
* Pregnant female
* Presence of ITP/autoimmune thrombocytopenia
* Immune platelet refractoriness responsive to treatment with IVIg or eculizumab, or other immunosuppressive therapy within the 3 preceding months. This is based on the wide variation in the duration therapeutic antibodies, with the upper limit frequently cited as 3 months.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Willy A Flegel, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared in de-identified format
Time Frame: After study completion
Access Criteria: Other researchers may access the data through Biomedical Translational Research Information System (BTRIS) database

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-CC-0005.html

RESULTS

PARTICIPANT FLOW:
Period: Block 1, Day 1
Arm/Group | Group A: LONG Then SHORT Transfusion | Group B: SHORT Then LONG Transfusion
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0
Period: Block 2, Day 2
Arm/Group | Group A: LONG Then SHORT Transfusion | Group B: SHORT Then LONG Transfusion
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0
Period: Block 3, Day 3
Arm/Group | Group A: LONG Then SHORT Transfusion | Group B: SHORT Then LONG Transfusion
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Participants: Subjects with thrombocytopenia (due to congenital causes, bone marrow failure, hematologic malignancies, and treatment-related) randomized to receive either LONG platelet transfusion (Transfused over 4-HOURS via infusion pump or gravity) or SHORT platelet transfusion (Transfused over 60-minutes via infusion pump or gravity) with follow up until six (6) hours for each transfusion for a combined total of 12 hours then cross over to receive subsequent intervention. Subjects may receive up to two further subsequent blocks (one per day) to be administered to a subject in alternating order, for a maximum number of three blocks per subject.
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Platelet Increment Area Under the Curve (AUC)
Description: The adjusted platelet increment area under the curve (AUC), obtained between 0-hours and 6-hours after start of the platelet transfusion. The AUC (i.e., AUC above the pretransfusion complete blood count (CBC) platelet count, minus the AUC below the pre-transfusion CBC's platelet count) determined by the 0-hour, 2-hour, 4-hour, and 6-hour CBC platelet concentrations, calculated using the trapezoid rule. Adjustment to the measured AUC done for the number of platelets transfused during the two transfusion periods (LONG and SHORT Transfusion durations) in one block.
Time Frame: 0-6 hours post transfusion
Population: Participants who completed at least one block of transfusion in the study
Measure: Mean (Standard Deviation); unit: platelets x 10^3 x min/uL
Groups:
- LONG Transfusion: Subjects with thrombocytopenia (due to congenital causes, bone marrow failure, hematologic malignancies, and treatment-related) randomized to receive LONG platelet transfusion (Transfused over 4-HOURS via infusion pump).
- SHORT Transfusion: Subjects with thrombocytopenia (due to congenital causes, bone marrow failure, hematologic malignancies, and treatment-related) randomized to receive SHORT platelet transfusion (Transfused within 60-minutes via infusion pump or gravity).
Arm/Group | LONG Transfusion | SHORT Transfusion
Number analyzed (Participants) | 2 | 2
platelets x 10^3 x min/uL | 1173.5 (669.2) | 746.9 (240.0)

2. Secondary Outcome: Participants With Bleeding During the Peri-transfusion Period
Description: The efficacy of continuous platelet infusion on bleeding outcomes was assessed by number of participants with bleeding grade 1 or higher, measured during the peri-transfusion period by daily hemostatic assessments using the World Health Organization (WHO) bleeding scale. The WHO Bleeding Scale is a standardized tool used to assess and grade the severity of bleeding from 0-4:
  Grade 0: No bleeding. Grade 1: Petechiae (small, pinpoint hemorrhages). Grade 2: Mild blood loss. Grade 3: Gross blood loss (visible blood loss). Grade 4: Debilitating blood loss (severe blood loss that causes weakness)
Time Frame: One day before the first Transfusion Block until one day after the last Transfusion Block; up to 5 days total
Population: Participants who completed at least one block of transfusion in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Long Transfusion | Short Transfusion
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 24 hours post platelet transfusion
Groups:
- LONG Transfusion: Subjects with thrombocytopenia (due to congenital causes, bone marrow failure, hematologic malignancies, and treatment-related) randomized to receive LONG platelet transfusion (Transfused over 4-HOURS via infusion pump or gravity) with follow up until 6 hours.
- SHORT Transfusion: Subjects with thrombocytopenia (due to congenital causes, bone marrow failure, hematologic malignancies, and treatment-related) randomized to receive SHORT platelet transfusion (Transfused over 60-minutes via infusion pump or gravity) with follow up until 6 hours.
Arm/Group | LONG Transfusion | SHORT Transfusion
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
Study was terminated due to recruitment issue

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-07): https://cdn.clinicaltrials.gov/large-docs/18/NCT03712618/Prot_SAP_000.pdf